CLINICAL TRIAL: NCT05529992
Title: A Multicenter, Open-label Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Velaglucerase Alfa in Chinese Subjects With Type 1 Gaucher Disease
Brief Title: A Study of Velaglucerase Alfa (VPRIV) in Chinese Children, Teenagers, and Adults With Type 1 Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-669-3001; 2022-002323-35 (EudraCT Number)
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Gaucher Disease
Keywords: VPRIV; Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Velaglucerase Alfa (VPRIV) (Experimental): Participants received VPRIV IV infusion at 60 units per kilogram (U/kg) body weight once every other week (EOW) for 60 (+10) minutes for up to 51 weeks.
  Interventions: Drug: Velaglucerase Alfa

INTERVENTIONS:
Drug: Velaglucerase Alfa — VPRIV intravenous infusion every other week for 60 minutes.
  Other Names: VPRIV

SUMMARY:
The main purpose of this study is to observe the side effects of VPRIV in participants with type 1 Gaucher disease who are either treatment-naïve (newly diagnosed) or who are currently being treated with enzyme replacement therapy (ERT).

Participants will receive VPRIV intravenously during the treatment period (up to 51 weeks), followed by the end-of-treatment (EOT) visit after 2 weeks.

DETAILED DESCRIPTION:
The drug being tested in this study is called Velaglucerase Alfa (VPRIV). VPRIV will be tested to treat participants with type 1 Gaucher disease. This study will look at the safety, efficacy and pharmacokinetics of VPRIV in the treatment of type 1 Gaucher disease.

The study will enroll approximately 20 participants with Gaucher disease. The study comprises a screening period (Day -21 through Day -4), baseline period (Day -3 through Day 0), treatment period (Week 1 to Week 51), and safety follow-up period. Participants will be assigned to the following drug administration:

• Velaglucerase Alfa (VPRIV)

Participants will receive VPRIV as intravenous (IV) infusion every other week from Week 1 through Week 51 during the Treatment Period. Percentage of participants with at least one serious treatment-emergent adverse event (TEAE) will be evaluated throughout the study.

This multi-center trial will be conducted in China. The overall time to participate in this study is approximately 59 weeks. Participants will make a safety follow-up telephone call or visit to the site after 30 (±7) days of the last infusion of the study drug.

ELIGIBILITY:
Inclusion:

* Has a documented, confirmed diagnosis of type 1 Gaucher disease based on the following, as determined by the investigator:

  1. Decreased glucocerebrosidase (GCB) activity level that is ≤30% of normal or
  2. Decreased GCB activity level that is >30% of normal, but with confirmation of genetic mutation test
* Is at least 2 years of age, inclusive, at screening
* Is naive to treatment for Gaucher disease (Has not received treatment for Gaucher disease [investigational or approved products] within the 12 months prior to screening) OR Is receiving or has recently received Imiglucerase ERT (Has received Imiglucerase treatment within the 12 months prior to screening and not within the 14 days prior to screening)
* Has Gaucher disease-related hematological abnormalities, defined as

  1. Hemoglobin levels of ≥1 g/dL below the lower limit of normal for their age and gender AND/OR
  2. A platelet count of <90 × 10^9/L below the lower limit of normal for their age and gender
* Has Gaucher disease-related viscera abnormalities, defined as the following:

  * Participant has at least moderate splenomegaly, assessed by palpation (2 to 3 cm below the left costal margin), or by abdominal radiology scan (magnetic resonance imaging [MRI] or computed tomography [CT] scan, with spleen volume >5 times normal) AND/OR
  * Participant has hepatomegaly, assessed by palpation or by abdominal radiology scan (MRI or CT scan); Participants who have undergone splenectomy must have satisfied these criteria for this study.

Exclusion:

* Has type 2 or 3 Gaucher disease or is suspected of having type 3 Gaucher disease as assessed by the investigator
* Has had a splenectomy or an active, clinically significant spleen infarction within the 12 months prior to screening
* Has received treatment with any investigational drug or device within 30 days prior to screening, or within 5 half-lives of that investigational product, whichever is greater; such treatment during the study will not be permitted
* Is currently receiving red blood cell growth factor (eg, erythropoietin), chronic systemic corticosteroids, or has been on such treatment within the 6 months prior to screening
* Presents with non-Gaucher disease related exacerbated anemia at screening
* Has experienced a severe (grade 3 or higher) infusion-related hypersensitivity reaction (anaphylactic or anaphylactoid reaction) to any ERT (approved or investigational)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- China (10):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/fba4cdf09dab492e?idFilter=%5B%22TAK-669-3001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites in China from 3 January 2023 to 5 August 2024.
Pre-assignment Details: Participants with a diagnosis of type 1 Gaucher disease were enrolled in this study to receive velaglucerase alfa (VPRIV) as intravenous (IV) infusion.
Groups:
- VPRIV: Participants received VPRIV IV infusion at 60 units per kilogram (U/kg) body weight once every other week (EOW) for 60 (+10) minutes up to Week 51.
Period: Overall Study
Arm/Group | VPRIV
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Set included all participants who signed the informed consent form (ICF) [and assent form, if applicable] and were eligible for the study based on the defined inclusion/exclusion criteria.
Groups:
- VPRIV: Participants received VPRIV IV infusion at 60 U/kg body weight once EOW for 60 (+10) minutes up to Week 51.
Arm/Group | VPRIV
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Serious Treatment-Emergent Adverse Event (TEAE)
Description: Adverse event(AE)=any untoward medical occurrence in clinical investigation participant administered a drug;it does not necessarily have to have causal relationship with this treatment. AE can therefore be any unfavorable&unintended sign (example,clinically significant abnormal laboratory value),symptom/disease temporally associated with use of drug whether or not it is considered related to drug. TEAE=any event emerging or manifesting at or after initiation of investigational product or any existing event that worsens in either intensity or frequency following exposure to investigational product. SAE=any untoward clinical manifestation of signs, symptoms, or outcomes(whether considered related to investigational product or not)&at any dose: results in death,is life-threatening,requires in-patient hospitalization/prolongation of hospitalization,results in persistent/significant disability/incapacity,results in congenital abnormality/birth defect,or is an important medical event.
Time Frame: Up to 56.2 weeks
Population: The Safety Set (SAF) included all participants in the ITT Set who received at least 1 dose of VPRIV.
Measure: Number; unit: percentage of participants
Arm/Group | VPRIV
Number analyzed (Participants) | 20
percentage of participants | 20

2. Secondary Outcome: Percentage of Participants With TEAEs
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory value), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. A TEAE is defined as any event emerging or manifesting at or after the initiation of the investigational product or any existing event that worsens in either intensity or frequency following exposure to the investigational product.
Time Frame: Up to 56.2 weeks
Population: The SAF included all participants in the ITT Set who received at least 1 dose of VPRIV.
Measure: Number; unit: percentage of participants
Arm/Group | VPRIV
Number analyzed (Participants) | 20
percentage of participants | 95

3. Secondary Outcome: Percentage of Participants With Infusion-related Reactions Reported as an Adverse Event
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory value), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. An infusion-related AE was defined as an AE that 1) began either during or within 12 hours after the start of the infusion and 2) was judged as possibly or probably related to the study treatment.
Time Frame: Up to 56.2 weeks
Population: The SAF included all participants in the ITT Set who received at least 1 dose of VPRIV.
Measure: Number; unit: percentage of participants
Arm/Group | VPRIV
Number analyzed (Participants) | 20
percentage of participants | 5

4. Secondary Outcome: Percentage of Participants With Development of Anti-VPRIV Antibodies and Neutralizing Antibodies at Week 53
Description: Percentages were rounded off to the nearest single decimal place.
Time Frame: Week 53
Population: The SAF included all participants in the ITT Set who received at least 1 dose of VPRIV. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | VPRIV
Number analyzed (Participants) | 19
percentage of participants
  Anti-VPRIV Antibodies | 15.8
  Neutralizing Antibodies | 10.5

5. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Assessments at Week 53
Description: Clinical laboratory assessments included hematology and serum chemistry. Any clinically significant changes in the clinical laboratory assessment values based on the investigator's interpretation were reported. Only categories with at least one participant with event are presented.
Time Frame: Week 53
Population: The SAF included all participants in the ITT Set who received at least 1 dose of VPRIV. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | VPRIV
Number analyzed (Participants) | 19
Participants
  Hematology: Erythrocytes Mean Corpuscular Hemoglobin Concentration | 2
  Hematology: Erythrocytes Mean Corpuscular Hemoglobin | 3
  Hematology: Erythrocytes Mean Corpuscular Volume | 2
  Hematology: Erythrocytes | 2
  Hematology: Hematocrit | 5
  Hematology: Hemoglobin | 4
  Hematology: Leukocytes | 2
  Hematology: Lymphocytes: number analyzed (Participants) | 17
  Hematology: Lymphocytes | 1
  Hematology: Monocytes: number analyzed (Participants) | 17
  Hematology: Monocytes | 1
  Hematology: Neutrophils: number analyzed (Participants) | 17
  Hematology: Neutrophils | 2
  Hematology: Platelets | 14
  Serum Chemistry: Bilirubin | 3
  Serum Chemistry: Ferritin | 5
  Serum Chemistry: Iron: number analyzed (Participants) | 17
  Serum Chemistry: Iron | 2

6. Secondary Outcome: Number of Participants With Abnormal Changes in Laboratory Assessments at Week 53: Urinalysis
Description: Any abnormal changes in the urinalysis assessment values based on the investigator's interpretation were reported. Urinalysis comprised of the following parameters: bilirubin, ketones, glucose, nitrite, occult blood, protein, and urobilinogen.
Time Frame: Week 53
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | VPRIV
Number analyzed (Participants) | 19
Participants
  Urinalysis: Bilirubin | 1
  Urinalysis: Ketones | 0
  Urinalysis: Glucose | 1
  Urinalysis: Nitrite | 1
  Urinalysis: Occult Blood: number analyzed (Participants) | 17
  Urinalysis: Occult Blood | 7
  Urinalysis: Protein | 3
  Urinalysis: Urobilinogen | 3

7. Secondary Outcome: Number of Participants With at Least One Abnormal Change in an Infusion Vital Sign Parameter at Week 53
Description: Participants with atleast 1 abnormal change (above or below normal) in an infusion vital sign parameter of pulse, temperature, respiratory rate,& blood pressure were reported. Normal ranges for each vital sign parameter were, pulse (beats per minutes [bpm]): 40-100(≥12 years old), 55-95(≥6 but <12 years old), 65-110(≥2 but <6 years old); body temperature(degree Celsius[˚C]): 36.5 to 37.2(all age groups),respiration rate(breaths/minutes):12-24(≥12 years old),12-22 (≥6 but <12 years old),20-30(≥2 but <6 years old);systolic blood pressure(BP) [millimeters of mercury{mm Hg}]: high: ≥140 (≥18 years old), ≥20+ 80+ 2*age(<18 years old), low: <90 (≥18 years old), < -20+ 80+ 2*age(<18 years old); diastolic BP(mm Hg):high:≥90 (≥18 years old), ≥20+ (80+2*age)*(2/3) (<18 years old) low: <50 (≥18 years old), < -20+ (80+2*age)*(2/3) (<18 years old). As per planned analysis,data was collected in a combined manner for all participants irrespective of age. Only non-zero categories are presented.
Time Frame: Week 53
Population: The SAF included all participants in the ITT Set who received at least 1 dose of VPRIV. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | VPRIV
Number analyzed (Participants) | 20
Participants
  Pulse: Above Normal | 15
  Body Temperature: Above Normal: number analyzed (Participants) | 18
  Body Temperature: Above Normal | 1
  Body Temperature: Below Normal: number analyzed (Participants) | 18
  Body Temperature: Below Normal | 18
  Respiratory Rate: Above Normal | 9
  Systolic BP: Above Normal | 11
  Systolic BP: Below Normal | 5
  Diastolic BP: Above Normal | 8
  Diastolic BP: Below Normal | 3

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Measurements at Week 53
Description: Participants with clinically significant changes in any ECG measurement, such as PR, QRS, QT, corrected QT intervals, and heart rate based on the investigator's interpretation were reported.
Time Frame: Week 53
Population: The SAF included all participants in the ITT Set who received at least 1 dose of VPRIV. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | VPRIV
Number analyzed (Participants) | 19
Participants | 1

9. Secondary Outcome: Change From Baseline to Week 53 in Hemoglobin Concentration
Time Frame: Baseline, Week 53
Population: The ITT Set included all participants who signed the ICF (and assent form, if applicable) and were eligible for the study based on the defined inclusion/exclusion criteria. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | VPRIV
Number analyzed (Participants) | 18
grams per deciliter (g/dL) | 2.34 (1.305)

10. Secondary Outcome: Change From Baseline to Week 53 in Platelet Count
Time Frame: Baseline, Week 53
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: platelets*10^9/liter
Arm/Group | VPRIV
Number analyzed (Participants) | 18
platelets*10^9/liter | 42.1 (27.68)

11. Secondary Outcome: Change From Baseline to Week 53 in Normalized Liver Volume
Description: Normalized liver volume was measured by abdominal magnetic resonance imaging (MRI) or computed tomography (CT) scan. Liver volume was normalized for percent body weight.
Time Frame: Baseline, Week 53
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of body weight (%BW)
Arm/Group | VPRIV
Number analyzed (Participants) | 19
percentage of body weight (%BW) | -1.11 (0.917)

12. Secondary Outcome: Change From Baseline to Week 53 in Normalized Spleen Volume
Description: Spleen volume was normalized for percent body weight.
Time Frame: Baseline, Week 53
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: % BW
Arm/Group | VPRIV
Number analyzed (Participants) | 19
% BW | -3.09 (1.627)

13. Secondary Outcome: Change From Baseline to Week 53 in 36-item Short Form General Health Survey (SF-36) Scores
Description: SF-36 Version 2 is a multipurpose, participant completed, short-form health survey with 36 questions that consists of an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures. Physical component summary (PCS) is mostly contributed by physical function (PF), role physical (RP), bodily pain (BP), and general health (GH). Mental component summary (MCS) is mostly contributed by mental health (MH), role emotional (RE), social function (SF), and vitality (VT). Each component on the SF-36 item health survey is scored from 0 (best) to 100 (worst). Total score ranges from 0-100 for each component summary (i.e., PCS and MCS), where higher scores are associated with less disability and better quality of life.
Time Frame: Baseline, Week 53
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VPRIV
Number analyzed (Participants) | 4
score on a scale
  Physical Component Summary | 7.015 (5.8464)
  Mental Component Summary | 2.858 (12.5103)

14. Secondary Outcome: Change From Baseline to Week 53 in Childhood Health Questionnaire-Parent Form 50 (CHQ-PF50) Scores
Description: The CHQ-PF-50 is a 50-item questionnaire to be completed by the parents or guardians of children between 5 and 18 years of age. The 50 questions measure 14 domains (global health, physical functioning, role/social limitations (emotional/behavioral and physical), bodily pain/discomfort, behavior, global behavior, mental health, self-esteem, general health perceptions, change in health, parental impact (emotional and time), family activities, and family cohesion) which were summarized as the physical and psychological summary scores. Each summary score was transformed and could range from 0 to 100, with higher score indicating better physical and psychosocial health. A positive change from Baseline indicates improved well-being.
Time Frame: Baseline, Week 53
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VPRIV
Number analyzed (Participants) | 15
score on a scale
  Physical Summary Score | -0.02 (12.745)
  Psychosocial Summary Score | 0.38 (11.462)

15. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for VPRIV at Week 1
Time Frame: Pre-dose and at multiple timepoints up to 120 minutes post-dose on Day 1 of Week 1
Population: The Pharmacokinetic (PK) Set included all naïve participants in the ITT set who received at least 1 dose of VPRIV and provided evaluable PK concentration data.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | VPRIV
Number analyzed (Participants) | 16
nanograms per milliliter (ng/mL) | 5220 (1610)

16. Secondary Outcome: Serum Concentration for VPRIV at Week 37
Time Frame: Within 3 minutes prior to the end of the 60-minute infusion at Week 37
Population: The PK Set included all naïve participants in the ITT set who received at least 1 dose of VPRIV and provided evaluable PK concentration data. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VPRIV
Number analyzed (Participants) | 15
ng/mL | 3450 (1390)

17. Secondary Outcome: Tmax: Time to Reach the Maximum Serum Concentration (Cmax) for VPRIV
Time Frame: Pre-dose and at multiple timepoints up to 120 minutes post-dose on Day 1 of Week 1
Population: The PK Set included all naïve participants in the ITT set who received at least 1 dose of VPRIV and provided evaluable PK concentration data.
Measure: Median (Full Range); unit: minutes (min)
Arm/Group | VPRIV
Number analyzed (Participants) | 16
minutes (min) | 49.00 [19.00 to 60.00]

18. Secondary Outcome: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for VPRIV
Description: ng*min/mL denotes nanograms*minutes per milliliter.
Time Frame: Pre-dose and at multiple timepoints up to 120 minutes post-dose on Day 1 of Week 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*min/mL
Arm/Group | VPRIV
Number analyzed (Participants) | 16
ng*min/mL | 235000 (85000)

19. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for VPRIV
Time Frame: Pre-dose and at multiple timepoints up to 120 minutes post-dose on Day 1 of Week 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: min
Arm/Group | VPRIV
Number analyzed (Participants) | 16
min | 10.12 (2.81)

20. Secondary Outcome: Oral Clearance (CL) for VPRIV
Description: mL/min/kg denotes milliliters per minutes per kilogram.
Time Frame: Pre-dose and at multiple timepoints up to 120 minutes post-dose on Day 1 of Week 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | VPRIV
Number analyzed (Participants) | 16
mL/min/kg | 7.27 (2.87)

21. Secondary Outcome: Apparent Steady-state Volume of Distribution (Vss) for VPRIV
Time Frame: Pre-dose and at multiple timepoints(up to 120 minutes post-dose on Day 1 of Week 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: milliliters per kilogram (mL/kg)
Arm/Group | VPRIV
Number analyzed (Participants) | 16
milliliters per kilogram (mL/kg) | 96.3 (52.0)

22. Secondary Outcome: Percent Change From Baseline to Week 53 in Biomarker: Plasma Chemokine [C-C Motif] Ligand 18
Time Frame: Baseline, Week 53
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | VPRIV
Number analyzed (Participants) | 19
percent change | -58.94 (14.339)

23. Secondary Outcome: Percent Change From Baseline to Week 53 in Biomarker: Glucopsychosine
Time Frame: Baseline, Week 53
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | VPRIV
Number analyzed (Participants) | 19
percent change | -63.88 (14.359)

ADVERSE EVENTS:
Time Frame: Up to 56.2 weeks
Description: The SAF included all participants in the ITT Set who received at least 1 dose of VPRIV.
Groups:
- Velaglucerase Alfa: Participants received VPRIV IV infusion at 60 U/kg body weight once EOW for 60 (+10) minutes up to Week 51.
Arm/Group | Velaglucerase Alfa
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Velaglucerase Alfa (N=20)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Splenic injury (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Velaglucerase Alfa (N=20)
Conjunctivitis (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Fall (Injury, poisoning and procedural complications) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Pneumonia (Infections and infestations) | 2
Pyrexia (General disorders) | 3
Supraventricular extrasystoles (Cardiac disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 14
Urinary occult blood positive (Investigations) | 2
Urinary tract infection (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT05529992/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT05529992/SAP_001.pdf